CLINICAL TRIAL: NCT02155283
Title: The Kyrobak Continuous Passive Motion Device for the Treatment of Chronic Low Back Pain: A Pilot Study
Brief Title: The Efficacy of the Kyrobak for Chronic Low Back Pain (LBP-2)
Acronym: LBP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiancy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBP-2
Record Dates: First submitted 2013-12-11; First posted 2014-06-04 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Mild-to-Moderate Chronic Low Back Pain; Continuous Passive Motion Devices
MeSH Terms: conditions — Low Back Pain | interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Continuous Passive Motion (Other): Single-arm; 3-week treatment plan using Kyrobak compared to baseline (before treatment)
  Interventions: Device: Continuous Passive Motion

INTERVENTIONS:
Device: Continuous Passive Motion — Daily self-treatments at home for 3 weeks, with up to three 10-minute treatment sessions per day
  Other Names: Kyrobak

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Kyrobak continuous passive motion home-use device in relieving low back pain, improving proprioception (balance and fall prevention) and improving the symmetry of muscle function on either side of the spine.

DETAILED DESCRIPTION:
The Kyrobak is an electrically operated, continuous passive motion device including a platform that performs angular oscillations. The Kyrobak is used at home as an aid to relieve mild-to-moderate low back pain.

The study is designed to evaluate the efficacy of daily home use of the Kyrobak for 3 weeks and to assess the sustained efficacy 1 week later.

The evaluation will include the level of pain using the numerical rating scale (NRS), Digital Posturography, Heart Rate Variability (HRV), Static Surface Electromyography (SEMG), a condition-specific low back pain disability status by the Oswestry Disability Index (ODI) and subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 or older
* Level of pain - mild to moderate low back pain (≤5 NRS pain)
* Chronic - symptoms must have been present for at least 12 weeks or more.
* Location - lower tip of scapula to back of pelvis
* Etiology - non-specific

Exclusion Criteria:

* Patients who have low back pain due to specific and known causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome (radiating nerve pain from the spine such as sciatica), cauda equinal syndrome (serious neurological disorder where the spinal nerve roots are compressed which can cause).
* Weight in excess of 265 lbs. (120.4 kg)
* Pregnant or breastfeeding
* Recent history of violent trauma
* History of previous back surgery
* Constant progressive, non-mechanical pain (no relief with bed rest)
* Chronic pain other than low back pain
* Past medical history of malignant tumor
* Has taken an investigational drug within the past 30 days prior to entering the study, or currently enrolled in another investigational study
* Mental disorder that would lead to difficulty in questionnaire completion
* Any litigation for low back pain
* Prolonged use of corticosteroids (i.e. used for 3 months or more)
* Present use of prescription pain medication (i.e. Percocet®, Oxycodone, Vicodin®, etc.)
* Physical disability that prevents the subject to lie down/get up
* Drug abuse, immunosuppression, HIV
* Any other condition which in the physician's opinion would make it unsafe for the subject to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Geanopulos, DC, Principal Investigator — New Heights Chiropractic
Locations (1):
- New Heights Chiropractic, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Continuous Passive Motion
Started | 16
Completed | 9
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Continuous Passive Motion
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.75 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Amount of Pain Determined by the NRS at the End of the 3-week Treatment Plan Compared to Baseline (Before Treatment)
Description: Pain level will be scored by the subject using the NRS on a 0 to 10 scale where 10 represents the highest level of pain and 0 represents no pain.
Time Frame: 3 weeks
Population: Completers per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Continuous Passive Motion
Number analyzed (Participants) | 9
units on a scale | -2.87 (1.71)

2. Secondary Outcome: Change in Proprioception and Vestibular Function.
Description: Gather information regarding:
  Balance and Fall Prevention using digital posturography
Time Frame: 3 weeks, 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change in Functional Health Status by ODI
Description: Functional health status will be determined by the ODI questionnaire completed by the subject (based upon answers from 10 multiple choice questions)
Time Frame: 3 weeks, 4 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in Symmetry of Muscle Function on Either Side of the Spine
Description: Gather information regarding:
  Symmetry of muscle function about the spine using static surface electromyography (SEMG)
Time Frame: 3 weeks, 4 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in Heart Rate Variability (and the Autonomic System)
Description: Gather information regarding:
  Autonomic nervous system activity by measuring heart rate variability (HRV).
Time Frame: 3 weeks, 4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Amount of Pain Determined by the NRS at the 1-week Follow-up After the End of the 3-week Treatment Plan Compared to Baseline (Before Treatment)
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Continuous Passive Motion
Number analyzed (Participants) | 9
units on a scale | -2.61 (1.51)

ADVERSE EVENTS:
Arm/Group | Treatment Continuous Passive Motion
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No